CLINICAL TRIAL: NCT04210583
Title: Multi-Polar RF and PEMF Technologies for the Treatment of Vaginal Laxity and for Treatment of the Mons Pubis and Labia for Improvement of Skin Laxity: 12-Month Safety and Efficacy
Brief Title: RF and PEMF for Treatment of Vaginal Laxity and Mons Pubis and Labia for Improvement of Skin Laxity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FE1019
Record Dates: First submitted 2019-12-13; First posted 2019-12-24 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Vulvovaginal Atrophy; Menopause; Menopause Surgical

STUDY DESIGN:
Intervention Model Description: 1. Long term safety of the Venus Fiore Fiore™ (MP)2 system in improving vaginal laxity and skin laxity of the mons pubis and labia.
     * Subject's assessment of discomfort and pain as measured by a 10 cm visual analog scale (VAS) at 12 months if treatment (optional) is provided.
     * Subjects experiencing a treatment-related adverse event (AE) at six-months and twelve-months post-treatment.
  2. Long term efficacy of the Venus Fiore Fiore™ (MP)2 system in improving vaginal laxity and skin laxity of the mons pubis and labia.
     * Improvement in vaginal laxity at six-months and twelve-months post-treatment compared to baseline as defined as a score >4 on the VLQ.
     * Improvement in FSFI mean score at six-months and twelve-months post-treatment compared to baseline.
Masking Description: 1. Long term safety of the Venus Fiore Fiore™ (MP)2 system in improving vaginal laxity and skin laxity of the mons pubis and labia.
     * Subject's assessment of discomfort and pain as measured by a 10 cm visual analog scale (VAS) at 12 months if treatment (optional) is provided.
     * Subjects experiencing a treatment-related adverse event (AE) at six-months and twelve-months post-treatment.
  2. Long term efficacy of the Venus Fiore Fiore™ (MP)2 system in improving vaginal laxity and skin laxity of the mons pubis and labia.
     * Improvement in vaginal laxity at six-months and twelve-months post-treatment compared to baseline as defined as a score >4 on the VLQ.
     * Improvement in FSFI mean score at six-months and twelve-months post-treatment compared to baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vulvovaginal Treatment (Experimental): At visit 1 -(6 months post treatment in the CS0716 study):
  AE assessment, VLQ, FSFI, GRAS and GAIS (optional), Vaginal pH and vaginal smear (optional),
  At Visit 2 (6 months post treatment in the CS0716 study):
  AE assessment, VLQ, FSFI, GRAS and GAIS (optional), Vaginal pH and vaginal smear (optional), Administer study treatment (optional: internal, mons pubis and/or labia treatment).
  Discomfort/pain 10 cm VAS, immediate response assessment (applicable only if treatment provided)
  Final AE follow-up 30 days post Visit 2 Treatment (if applicable): AE assessment (applicable only if treatment provided at Visit 2 in the FE1019 study).
  Interventions: Device: Vulvovaginal Treatment

INTERVENTIONS:
Device: Vulvovaginal Treatment — Device model(s) - Venus Fiore™ Device settings and programming internal applicator - 42°C - 45°C Temperature output via automatic temperature control (ATC) (optional treatment).
  Duration of exposure and frequency of exposure with internal applicator - one treatment for 12-15 minutes at 12 months (optional treatment).
  Device settings and programming external mons pubis and labia applicators - 10-35% output (optional treatment).
  Duration of exposure and frequency of exposure external applicators - one treament for 15 minutes for the mons pubis, 10 minutes for labia at 12 months (optional treatment).

SUMMARY:
Twelve month extension of a previous study of Multi-Polar RF and PEMF technologies for the treatment of vaginal laxity and for the treatment of the mons pubis and labia for improvement in skin laxity. The study will enroll up to 50 subjects who completed the Venus Fiore CS0716 study for the treatment of vaginal laxity and treatment of the mons pubis and labia for improvement in skin laxity. Subjects will be followed up at least six and twelve months post-treatment. Analysis will be performed on all subjects who complete the six-month and twelve month follow-up visits.

DETAILED DESCRIPTION:
Traditional non-surgical treatments to treat vaginal laxity include Kegel exercises or pelvic floor therapy with electrical stimulation of the vaginal musculature to promote muscle strength. Although surgery to tighten the vaginal introitus has been used, pain at the incision site leading to dyspareunia, sometimes for months, limits its use. Surgery is also recommended to reduce protuberant mons pubis and the outer labial lips of the labia majora. Most often, the mons pubis has been treated by fat reduction, either by liposuction or open excision along with a pubic skin lift. Surgery to reduce the excess skin of the labia majora tends to be avoided due to a lack of operative techniques and a fear of creating sexual dysfunction. Development of alternative methods of treatment, avoiding the usual surgical complications is warranted.

The use of non-ablative radiofrequency (RF) therapy has been used previously for the external and internal female genitalia without incident or complications. The use of Multi-Polar RF and PEMF technology was already demonstrated to be safe and efficient in delivering heat to the tissue. A previous study investigated the safety and efficacy of combining these technologies for the treatment of vaginal laxity and in the treatment of the mons pubis and labia for the improvement in skin laxity at four-months post-treatment. Efficacy and safety was confirmed up to 4-months post-treatment. (Venus FioreTM CS0716 study, unpublished raw data). However, the durability of the treatment is not known.

This study will investigate whether Multi-Polar RF and PEMF technologies for the treatment of vaginal laxity and for the treatment of the mons pubis and labia is safe and efficacious at six-months and twelve-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed at least two treatments in the Venus Fiore™ CS0716 study and are at least 6 months post Fiore™ treatment.
2. Able to read, understand and voluntarily provide written Informed Consent.
3. Able and willing to comply with the treatment/follow-up schedule and requirements.
4. Sexual active and in a monogamous relationship

Exclusion Criteria:

1. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
2. Having a permanent implant in the treatment area.
3. Prior use of collagen, fat injections and/or other methods of skin augmentation (enhancement with injected or implanted material) in the treatment areaduring the course of the study.
4. Use of retinoids such as oral Isotretinoin (Accutane®) during the course of the study.
5. Any other surgery in treated area within 12 months of initial treatment or during the course of the study.
6. Open laceration, abrasion or bleeding of any sort on the areas to be treated.
7. Active sexual transmitted disease (STD) (e.g. genital Herpes Simplex, condylomata) or vaginosis.
8. Chronic vulvar pain or vulvar dystrophy.
9. Use of immunosuppressive medications, including corticosteroids, during the course of the study.
10. Having any form of active cancer at the time of enrollment and during the course of the study.
11. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Investigator would interfere with the study, or healing process.
12. Participation in a study of another device or drug within 1 month prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria.
13. Evidence of active substance or alcohol abuse.
14. Having any stage 3-4 cystocele, rectocele, enterocele paravaginal defect or major pelvic organ prolapse beyond the hymenal ring.
15. Unstable dosages of medications such as antihypertensives or use of psychotropics that are known to affect sexuality.
16. Skin piercing in the treatment area.
17. Tattoos in the treatment area.
18. Prior procedure in the treatment area with laser or other device during the course of the study.
19. Use of an intrauterine device during the course of the study.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible Females that have completed at least two treatments in the Venus Fiore™ CS0716 study and are at least 6 months post Fiore™ treatment.
Enrollment: 10 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Long term safety (Follow-up for any AEs) of the Venus Fiore Fiore™ (MP)2 system in vaginal laxity and skin laxity of the mons pubis and labia. | 6 months
  AE assessment VLQ, FSFI, GRAS and GAIS (optional) Vaginal pH and vaginal smear (optional) Discomfort/pain 10 cm VAS, immediate response assessment (applicable only if treatment provided)

SECONDARY OUTCOMES:
long term safety of the Venus Fiore Fiore™ (MP)2 system in improving vaginal laxity and skin laxity of the mons pubis and labia. | 12 months
  AE assessment VLQ, FSFI, GRAS and GAIS (optional) Vaginal pH and vaginal smear (optional) Administer study treatment (optional: internal, mons pubis and/or labia treatment) Discomfort/pain 10 cm VAS, immediate response assessment (applicable only if treatment provided)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Gronski, Study Director — Venus Concept
Locations (1):
- Dr. George Arnold, Markham, Ontario, Canada